CLINICAL TRIAL: NCT03847584
Title: Recruiting Participants With Low Socioeconomic Status in the NutriQuébec Study: Using Survey to Explore Their Beliefs, Preferences and Concerns
Brief Title: Using Survey to Explore Perceptions of Adults With Low Socioeconomic Status Regarding the NutriQuébec Study
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-042 A-2/10-09-2018
Record Dates: First submitted 2019-01-10; First posted 2019-02-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Survey
Keywords: Low socioeconomic status population; Web-based prospective cohort study; Survey; Recruitment; Attitude; Subjective norms; Perceived behavioural control; Intention
MeSH Terms: conditions — Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults-low socioeconomic status: Survey completed by adults with low socioeconomic status
  Interventions: Other: Survey
- Adults-middle/high socioeconomic status: Survey completed by adults with middle/high socioeconomic status
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The survey is based on the Theory of Planned Behaviour and assesses intention to participate in NutriQuébec as well as attitude, subjective norm, and perceived behavioural control. The salient beliefs underlying the determinants of individual's intention to participate in the NutriQuébec study most frequently cited in the focus groups (from a preliminary elicitation study: 2018-042 A-1/18-05-2018) were used to develop the survey questions. The survey also assesses the preferences regarding the recruitment. Sociodemographic questions are also asked.

SUMMARY:
Populations with low socioeconomic status (SES) are more likely to develop diseases across lifespan and are frequently underrepresented in large cohort studies. The aim of this study is to examine beliefs, preferences and concerns towards participating in an e-cohort prospective study on nutrition (NutriQuébec) among this population.

A cross-sectional survey will be completed by 418 adults in the Province of Québec (Canada), including individuals with low SES (high school or less and gross annual household income < $55,000 canadian). The survey is based on the Theory of Planned Behaviour and assesses intention to participate in NutriQuébec as well as attitude, subjective norm, and perceived behavioural control. The survey also assesses preferences regarding the recruitment.

DETAILED DESCRIPTION:
A cross-sectional survey will be completed by 418 participants from several administrative regions of Québec (Canada). A special effort will be made to recruit men and women with low socioeconomic status (SES), but without rejecting adults from middle/high SES. First, 325 adults from low SES (high school or less and gross annual household income < $55,000 canadian) and from several administrative regions of Québec will be identified by a survey firm. In addition, an e-mail mailing list from the Institute of Nutrition and Functional Food (INAF, Laval University) will be used to distribute the recruitment ad to complete our sample (n=93 from all SES).

The survey is based on the Theory of Planned Behaviour and assesses intention to participate in NutriQuébec as well as attitude, subjective norm, and perceived behavioural control. The salient beliefs underlying the determinants of individual's intention to participate in the NutriQuébec study most frequently cited in the focus groups (from a preliminary elicitation study: 2018-042 A-1/18-05-2018) were used to develop the survey questions. The survey also assesses the preferences regarding the recruitment. Sociodemographic questions are also asked.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older)
* Living in the province of Québec
* Have access to the Internet and have an active email address
* Be able to answer questionnaires in French

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with low/middle/high socioeconomic status
Sampling Method: Non-Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
The intention to participate to the NutriQuébec study will be assessed by a questionnaire based on the Theory of Planned Behaviour. | Baseline
  Intention will be calculated as the mean of three questions on a five point bipolar Likert scale. The three questions are: 1) I intend to participate in the NutriQuébec study : 1=very unlikely, 2=rather unlikely, 3=neither likely nor unlikely, 4=rather likely, 5=very likely; 2) The chances that I participate in the NutriQuébec study are : 1=very small, 2=rather small, 3=neither high nor small, 4=rather high, 5=very high; 3) I will participate in the NutriQuébec study: 1=very unlikely, 2=rather unlikely, 3=neither likely nor unlikely, 4=rather likely, 5=very likely). Thus, the mean score for intention ranges from 1 to 5, with higher values reflecting a greater likelihood for participation in the NutriQuébec study.
The attitude related to a hypothetical participation in the NutriQuébec study will be assessed by a questionnaire based on the Theory of Planned Behaviour. | Baseline
  The attitude will be calculated as the mean of three questions on a five point bipolar Likert scale. The three questions are: 1) For me, participating in the NutriQuébec study would be...: 1=very unpleasant, 2=rather unpleasant, 3=neither pleasant nor unpleasant, 4=rather pleasant, 5=very pleasant; 2) For me, participating in the NutriQuébec study would be...: 1=very useless, 2=rather useless, 3=neither useful nor useless, 4=rather useful, 5=very useful; 3) For me, participating in the NutriQuébec study would be…: 1=very unsatisfactory, 2=rather unsatisfactory, 3=neither satisfactory nor unsatisfactory, 4=rather satisfactory, 5=very satisfactory. Thus, the mean score for attitude ranges from 1 to 5, with higher values reflecting a more positive attitude towards a participation in the NutriQuébec study.
The subjective norm related to a hypothetical participation in the NutriQuébec study will be assessed by a questionnaire based on the Theory of Planned Behaviour. | Baseline
  The subjective norm will be calculated as the mean of three questions on a five point bipolar Likert scale. The three questions are: 1) The people most important to me might think that I should participate in the NutriQuébec study:1=very unlikely, 2=rather unlikely, 3=neither likely nor unlikely, 4=rather likely, 5=very likely; 2) Many people I know may be interested in participating in the NutriQuébec study: 1=very unlikely, 2=rather unlikely, 3=neither likely nor unlikely, 4=rather likely, 5=very likely; 3) If I participated in the NutriQuébec study, most people who are important to me could...: 1= strongly disapprove, 2= slightly disapprove, 3=neither approve nor disapprove, 4= slightly approve, 5=strongly approve. Thus, the mean score for the subjective norm ranges from 1 to 5, with higher values representing perceptions that important others expect the participant to participating in the NutriQuébec study.
The perceived behavioural control related to a hypothetical participation in the NutriQuébec study will be assessed by a questionnaire based on the Theory of Planned Behaviour. | Baseline
  The perceived behavioural control will be calculated by the mean of three questions on a five point bipolar Likert scale. The three questions are: 1) I feel able to participate in the NutriQuébec study: 1=very unlikely, 2=rather unlikely, 3=neither likely nor unlikely, 4=rather likely, 5=very likely; 2) I am confident that I can overcome any obstacles that may prevent me from participating in the NutriQuébec study: 1=very unlikely, 2=rather unlikely, 3=neither likely nor unlikely, 4=rather likely, 5=very likely; 3) For me, participating in the NutriQuébec study would be....: 1=very difficult, 2=rather difficult, 3=neither easy nor difficult, 4=rather easy, 5=very easy. Thus, the mean score for the perceived behavioural control ranges from 1 to 5, with higher values representing a greater perceived behavioural control towards a participation in the NutriQuébec study.
The determinants to the intention to participate to the NutriQuébec study will be assessed by a questionnaire based on the Theory of Planned Behaviour. | Baseline
  Determinants to the intention to participate in the NutriQuébec study will be identified with a multiple linear regression using constructs that will be found significant in influencing the intention to participate in the NutriQuébec study (e.g. attitude, subjective norm, perceived behavioural control).

SECONDARY OUTCOMES:
The preferences about the recruitment in the NutriQuébec study will be assessed by a questionnaire | Baseline
  The preferences about the recruitment in the NutriQuébec study will be assessed by a questionnaire. The question is: By which means of communication would advertising about the NutriQuébec study be most likely to capture your attention?: 1=Television, 2=Social networks (Facebook, Instagram, YouTube, etc.), 3=The Internet (other than social networks), 4=Newspapers, 5=Posters in public places (hospitals, community centres, etc.), 6=Flyers, 7=Postal mail, 8=None.

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Canada